CLINICAL TRIAL: NCT02698176
Title: A Phase IB Dose Exploration Trial With MK-8628, a Small Molecule Inhibitor of the Bromodomain and Extra-Terminal (BET) Proteins, in Subjects With Selected Advanced Solid Tumors
Brief Title: A Dose Exploration Study With Birabresib (MK-8628) in Participants With Selected Advanced Solid Tumors (MK-8628-006)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to limited efficacy and not due to safety reasons.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8628-006; MK-8628-006 (Other: Merck Protocol Number); 2015-005488-18 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: NUT Midline Carcinoma (NMC); Triple Negative Breast Cancer (TNBC); Non-small Cell Lung Cancer (NSCLC); Castration-resistant Prostate Cancer (CRPC)
Keywords: OTX015; MK-8628
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — OTX015

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Birabresib 20 mg CRPC Cohort-Part A (Experimental): Participants in the CRPC cohort in Part A of the study received birabresib 20 mg orally (PO), twice a day (BID), in a fasted state for 21 consecutive days per cycle. Participants received birabresib in continuous cycles up to 24 months.
  Interventions: Drug: Birabresib
- Birabresib 20 mg NMC Cohort-Part A (Experimental): Participants in the NMC cohort in Part A of the study received birabresib 20 mg PO, BID, in a fasted state for 21 consecutive days per cycle. Participants received birabresib in continuous cycles up to 24 months.
  Interventions: Drug: Birabresib
- Birabresib 20 mg TNBC Cohort-Part A (Experimental): Participants in the TNBC cohort in Part A of the study received birabresib 20 mg PO, BID, in a fasted state for 21 consecutive days per cycle. Participants received birabresib in continuous cycles up to 24 months.
  Interventions: Drug: Birabresib
- NMC Cohort-Part B (Experimental): Participants (up to 30) in Part B will receive birabresib at one dose level below the dose currently being administered in Part A of the study. Once the recommended Phase 2 dose (RP2D) from Part A is established, participants in Part B will receive birabresib at the RP2D. Participants will continue receiving birabresib at an assigned/adjusted dose level for continuous cycles up to 24 months.
  Interventions: Drug: Birabresib

INTERVENTIONS:
Drug: Birabresib — Administered as an oral capsule in a fasted state
  Other Names: OTX015; MK-8628

SUMMARY:
This is a study to determine the recommended dose of birabresib (MK-8628)(formerly known as OTX015) for further studies in participants with advanced nuclear protein in testis (NUT) midline carcinoma (NMC), triple negative breast cancer (TNBC), non-small cell lung cancer (NSCLC), or castration-resistant prostate cancer (CRPC). This is a two-part parallel study: Part A will establish the recommended dose by evaluating dose limiting toxicity (DLT), safety, discontinuation, and early efficacy and Part B will enroll participants with NMC only and will evaluate safety and efficacy in this population.

DETAILED DESCRIPTION:
The sponsor decided to terminate the program after evaluation of safety and efficacy data at the dose levels tested (Part A). The decision to discontinue the birabresib program was based on limited efficacy signals and was not due to safety-related concerns. No participants entered or were treated in Part B of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age for NSCLC, TNBC, and CRPC
* Males and females ≥16 years of age for NMC
* Diagnosis of one of the following advanced solid tumors for which standard therapy either does not exist or has proven ineffective, intolerable or inacceptable for the participant: NMC;TNBC; NSCLC; or CRPC
* Have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. CRPC participants may be enrolled with objective evidence of disease as per Prostate Cancer Working Group (PCWG2) criteria
* Life expectancy ≥3 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
* Have an interval of ≥3 weeks (or ≥2 weeks for NMC participants) since chemotherapy (≥6 weeks for nitrosoureas or mitomycin C), immunotherapy, hormone therapy or any other anticancer therapy or surgical intervention resection, or ≥3 half-lives for monoclonal antibodies, or ≥5 half-lives for other non-cytotoxic agents (whichever is longer)
* CRPC participants must maintain ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue, antagonist or orchiectomy providing serum testosterone is <50 ng/dL (<1.7 nmol/L)
* Participants receiving bisphosphonate or denosumab therapy must be on stable doses for at least 4 weeks before start of study therapy
* Females must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours of study start)
* Females of childbearing potential and male participants must agree to use adequate contraception starting with the first dose of trial treatment through 90 days after the last dose of study medication

Exclusion Criteria:

* Has inability to swallow oral medications or presence of a gastrointestinal disorder (e.g. malabsorption) deemed to jeopardize intestinal absorption of birabresib
* Has persistent grade >1 clinically significant toxicities related to prior antineoplastic therapies (except for alopecia). Stable sensory neuropathy ≤ grade 2 National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 is accepted
* Known primary central nervous system (CNS) malignancy or symptomatic or untreated CNS metastases. Treated and stable CNS metastases are allowed.
* History of prior or concomitant malignancies within 3 years of study start
* Have other serious illness or medical condition, such as active infection, unresolved bowel obstruction, psychiatric disorders, or cerebrovascular accident within 1 year of study start
* Known human immunodeficiency virus (HIV) and/or active Hepatitis B or C infections
* Have one of the following cardiac-related conditions: Congestive heart failure or angina pectoris (except if medically controlled); myocardial infarction (within 1 year of study start); uncontrolled hypertension; or uncontrolled arrhythmias
* Other concomitant anticancer treatment
* Participation in another clinical trial or treatment with any investigational drug (excluding anticancer treatments) within 30 days of study start
* Concomitant therapy with strong CYP3A4 inhibitors or inducers
* Therapeutic anticoagulation (e.g. warfarin, heparin, etc.) must be stopped at least 7 days prior to the first dose of birabresib. Low-dose low molecular weight heparin (LMWH) is permitted
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a dose-escalating study in participants with advanced or metastatic non-small cell lung cancer (NSCLC), triple negative breast cancer (TNBC), castration-resistant prostate cancer (CRPC), or nuclear protein in testis (NUT) midline carcinoma (NMC) for which standard therapy does not exist, proven ineffective, intolerable, or unacceptable.
Pre-assignment Details: Participants with CRPC, NMC, and TNBC, as defined in the entry criteria, were enrolled; no participants with NSCLC were enrolled. All participants had a Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤1 and 76.9% of participants had 2 or more prior lines of therapy. No participants were enrolled in Part B of the study.
Groups:
- MK-8628 20 mg CRPC Cohort-Part A: Participants in the CRPC cohort in Part A of the study received MK-8628 20 mg orally (PO), twice a day (BID), in a fasted state for 21 consecutive days per cycle. Participants received MK-8628 in continuous cycles up to 24 months.
- MK-8628 20 mg NMC Cohort-Part A: Participants in the NMC cohort in Part A of the study received MK-8628 20 mg PO, BID, in a fasted state for 21 consecutive days per cycle. Participants received MK-8628 in continuous cycles up to 24 months.
- MK-8628 20 mg TNBC Cohort-Part A: Participants in the TNBC cohort in Part A of the study received MK-8628 20 mg PO, BID, in a fasted state for 21 consecutive days per cycle. Participants received MK-8628 in continuous cycles up to 24 months.
- NMC Cohort-Part B: Participants (up to 30) in Part B were to receive MK-8628 at one dose level below the dose that was currently being administered in the escalation portion of Part A of the study. Once the recommended Phase 2 dose (RP2D) from Part A was established, participants in Part B were to receive MK-8628 at the RP2D. Participants were to continue receiving MK-8628 at an assigned/adjusted dose level for continuous cycles up to 24 months.
Period: Overall Study
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Started | 9 | 3 | 1 | 0 (No participants were enrolled in Part B.)
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 3 | 1 | 0
Not completed — Progressive disease | 4 | 3 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Clinical progression | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-8628 20 mg CRPC Cohort-Part A: Participants in the CRPC cohort in Part A of the study received MK-8628 20 mg PO, BID, in a fasted state for 21 consecutive days per cycle. Participants received MK-8628 in continuous cycles up to 24 months.
- Total: Total of all reporting groups
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | Total
Number analyzed (Participants) | 9 | 3 | 1 | 13
Age, Continuous [Mean (Full Range); unit: Years] | 71.2 [67 to 81] | 42.7 [30 to 67] | 66.0 [66 to 66] | 64.2 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 9 | 2 | 0 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 3 | 1 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT) During Cycle 1
Description: A DLT was any of the following deemed drug related (DR) by investigator: Grade (G)4 hematologic toxicity lasting ≥7 days except thrombocytopenia; G4 thrombocytopenia; G3 thrombocytopenia with bleeding; G3 or 4 febrile neutropenia. G4 non-hematologic (NH) toxicity (not laboratory); G3 NH toxicity (not laboratory), nausea, vomiting, or diarrhea lasting >3 days despite supportive care; G3 or 4 NH laboratory abnormality requiring medical intervention, hospitalization, or persisting >1 week; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >8X Upper Limit of Normal(ULN); ALT or AST >5XULN for >2 weeks; ALT or AST >3XULN and total bilirubin >2XULN or international normalization ratio >1.5; ALT or AST >3XULN with fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (>5%); DR adverse event leading to discontinuation or >20% missed planned doses in Cycle 1; DR toxicity causing >2 week delay in starting Cycle 2; or G5 toxicity.
Time Frame: From time of first dose up to the end of the first cycle (up to 21 days)
Population: Participants in Part A of the study that received at least 85% of the planned MK-8628 20 mg dose (18 days) or experienced a DLT during the first 21-day cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A
Number analyzed (Participants) | 9 | 3 | 1
Participants | 2 | 1 | 0
Statistical Analysis 1: Comparison: MK-8628 20 mg CRPC Cohort-Part A vs MK-8628 20 mg NMC Cohort-Part A vs MK-8628 20 mg TNBC Cohort-Part A; Test type: Other; Estimation of DLT Rate = 0.25, 80% CI 2-sided [0.121 to 0.418] — Point estimate and 2-sided 80% Bayesian credible interval for DLT rate estimated for the total number of participants from all 3 cohorts (CRPC+NMC+TNBC) that were evaluable for DLT analysis based on a non-informative prior distribution of Beta (1,1)

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: From time of first dose until the end of the 30-day follow-up (up to 25 months)
Population: Participants in Part A of the study that received at least 1 dose of MK-8628 20 mg. No participants were enrolled in Part B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Number analyzed (Participants) | 9 | 3 | 1 | 0
Participants | 9 | 3 | 1 |

3. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: From time of first dose until the end of treatment (up to 24 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Number analyzed (Participants) | 9 | 3 | 1 | 0
Participants | 2 | 0 | 0 |

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1) and lack of progression according to the guidelines for prostate cancer endpoints developed by Prostate Cancer Clinical Trials Working Group (PCWG) 2 as assessed by investigator radiologic review. The number of participants who achieved a CR or PR is presented.
Time Frame: Assessed every 6 weeks from time of first dose until disease progression (up to 24 months)
Population: Participants in Part A of the study who received at least one dose of MK-8628 20 mg. No participants were enrolled in Part B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Number analyzed (Participants) | 9 | 3 | 1 | 0
Participants | 0 | 0 | 0 |

5. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated CR or PR, DOR was defined as the time from first documented evidence of CR or PR per RECIST 1.1 until disease progression per RECIST 1.1 and PCWG2 or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression per RECIST 1.1. Per PCWG2, progressive disease was defined as a confirmed increase of at least two new lesions on a bone scan. DOR assessments were assessed by investigator radiologic review. The DOR for all participants who experienced a CR or PR is presented.
Time Frame: Assessed every 6 weeks from time of first dose until disease progression (up to 24 months)
Population: Participants in Part A of the study who received at least one dose of MK-8628 20 mg. No participants were enrolled in Part B of the study. Since no participants experienced a CR or PR, DOR could not be calculated.
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the number of subjects with CR, PR, or stable disease (SD) as assessed by investigator radiologic review according to RECIST version 1.1 and PCWG2. CR: defined as disappearance of all target and all non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than <10 mm per RECIST 1.1. PR: defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters along with absence of new lesions and disease progression in non-target lesions per RECIST 1.1. SD: defined as, neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study per RECIST 1.1 and lack of a confirmed increase of at least two new lesions on a bone scan per PCWG2. The number of participants who experienced DCR is presented.
Time Frame: Assessed every 6 weeks from time of first dose until disease progression (up to 24 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A | NMC Cohort-Part B
Number analyzed (Participants) | 9 | 3 | 1 | 0
Participants | 6 | 0 | 0 |

7. Secondary Outcome: Observed Maximum Concentration (Cmax) of MK-8628
Description: Blood samples were obtained at specified time points for the pharmacokinetic (PK) analysis of Cmax of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The Cmax of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: Total number of participants from all 3 cohorts (CRPC+NMC+TNBC) in Part A of the study that received at least 1 dose of MK-8628 20 mg and had data available for the PK parameter being analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MK-8628 20 mg PK Cohort: Total number of participants from all 3 cohorts (CRPC+NMC+TNBC) in Part A of the study that received at least 1 dose of MK-8628 20 mg PO, BID, in a fasted state.
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
ng/mL | 355 (157)

8. Secondary Outcome: Observed Minimum Concentration (Cmin) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Cmin of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The Cmin of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
ng/mL | 111 (45.9)

9. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Tmax of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The Tmax of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
hours | 2.25 [1.00 to 3.25]

10. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of t1/2 of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The t1/2 of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
hours | 6.17 (1.17)

11. Secondary Outcome: Apparent Total Body Clearance (CL/F) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Cl/F of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The Cl/F of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
Liters/hour | 6.44 (2.23)

12. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of MK-8628
Description: Blood samples were obtained at specified time points for the PK analysis of Vz/F of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The Vz/F of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | MK-8628 20 mg PK Cohort
Number analyzed (Participants) | 13
Liters | 55.0 (15.3)

13. Secondary Outcome: Area Under the Concentration-time Curve of MK-8628 From Time 0 to Infinity (AUC 0-∞)
Description: Blood samples were obtained at specified time points for the PK analysis of AUC 0-∞ of MK-8628. MK-8628 concentrations were analyzed using ultra-performance liquid chromatography coupled with a tandem mass spectrometry. The AUC 0-∞ of MK-8628 after oral administration is presented.
Time Frame: Cycle1/Day 1: predose, 20 minutes, 1 hour, 2.25 hours (hrs), 3.25 hrs, 8 hrs, and 12 hrs postdose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours•ng/mL
Groups:
- MK-8628 20 mg DLT Cohort: Total number of participants from all 3 cohorts (CRPC+NMC+TNBC) in Part A of the study that received at least 1 dose of MK-8628 20 mg PO, BID, in a fasted state.
Arm/Group | MK-8628 20 mg DLT Cohort
Number analyzed (Participants) | 13
hours•ng/mL | 3520 (1410)

ADVERSE EVENTS:
Time Frame: From time of first dose until the end of the 30-day follow-up (up to 25 months)
Description: The safety population consisted of all participants who received at least one dose of study treatment.
Arm/Group | MK-8628 20 mg CRPC Cohort-Part A | MK-8628 20 mg NMC Cohort-Part A | MK-8628 20 mg TNBC Cohort-Part A
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 20 mg CRPC Cohort-Part A (N=9) | MK-8628 20 mg NMC Cohort-Part A (N=3) | MK-8628 20 mg TNBC Cohort-Part A (N=1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 20 mg CRPC Cohort-Part A (N=9) | MK-8628 20 mg NMC Cohort-Part A (N=3) | MK-8628 20 mg TNBC Cohort-Part A (N=1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (7) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to limited efficacy and not due to safety reasons. Due to limited PK sampling for t1/2, caution must be exercised when interpreting the results of t1/2, CL/F, and AUC 0-∞ values.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/76/NCT02698176/Prot_SAP_000.pdf